CLINICAL TRIAL: NCT01996410
Title: The Efficacy of Acupuncture in Treating Chemotherapy Side Effects in Breast Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, John Elliott, Research Specialist- Medical Education, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OH1-13-00465
Record Dates: First submitted 2013-11-11; First posted 2013-11-27 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer Stages I Through III
Keywords: Breast Cancer; Acupuncture; Taxol; Cytoxan; Adriamycin; Taxotere; Carboplatin; Perjeta; Chemotherapy; Chemotherapy-induced nausea, vomiting; Chemotherapy-induced peripheral neuropathy; Adriamycin (60 mg/m2), Cytoxan (600 mg/m2), Taxol (175 mg/m2); Adriamycin (60 mg/m2), Cytoxan (600 mg/m2), Taxol (80 g/m2); Taxotere (75mg/m2), Cytoxan (600 mg/m2); Taxotere (75 mg/m2), Carboplatin (AUC 6), Perjeta (840 mg loading fixed dose)
MeSH Terms: conditions — Breast Neoplasms; Vomiting | interventions — Acupuncture Therapy

ARMS (8):
- Chemotherapy 1 Acupuncture (Active Comparator): Chemotherapy 1: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) concurrently on day 1 every 2 weeks for 4 cycles followed by Taxol (175mg/m2) on day 1 every 2 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every treatment for a total of 8 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 8 MDASI forms.
  Interventions: Device: Acupuncture
- Chemotherapy 2 Acupuncture (Active Comparator): Chemotherapy 2: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) on day 1 every 2 weeks for 4 cycles followed by Taxol (80mg/m2) on day 1 weekly for 12 cycles. Patients who randomize to the experimental ("acupuncture") group will undergo acupuncture the morning of every treatment day of the adriamycin/cytoxan cycles; they will receive acupuncture for every third Taxol treatment, beginning with the first treatment. They will receive a total of 8 acupuncture sessions: 4 with the adriamycin/cytoxan cycles and 4 with the Taxol cycles. Both groups will fill out MDASI on day 3 (+/- 1 days) of each Adriamycin/Cytoxan cycle; they will also fill out the MDASI on day 3 (+/- 1 days) of every third Taxol treatment for a total of 8 MDASI forms.
  Interventions: Device: Acupuncture
- Chemotherapy 3 Acupuncture (Active Comparator): Chemotherapy 3: In the adjuvant setting- This group will receive Taxotere (75mg/m2) and Cytoxan (600 mg/m2) on day 1 every 3 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Cytoxan for a total of 4 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 4 MDASI forms.
  Interventions: Device: Acupuncture
- Chemotherapy 4 Acupuncture (Active Comparator): Chemotherapy 4: In the neoadjuvant setting- This group will receive Taxotere (75 mg/m2), Carboplatin (AUC 6), Perjeta (840 mg loading fixed dose, followed by 420 mg maintenance fixed dose) day 1 every 3 weeks for 6 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Carboplatin/Perjeta treatment for a total of 6 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 6 MDASI forms.
  Interventions: Device: Acupuncture
- Chemotherapy 1 No Acupuncture (No Intervention): Chemotherapy 1: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) concurrently on day 1 every 2 weeks for 4 cycles followed by Taxol (175mg/m2) on day 1 every 2 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every treatment for a total of 8 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 8 MDASI forms.
- Chemotherapy 2 No Acupuncture (No Intervention): Chemotherapy 2: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) on day 1 every 2 weeks for 4 cycles followed by Taxol (80mg/m2) on day 1 weekly for 12 cycles. Patients who randomize to the experimental ("acupuncture") group will undergo acupuncture the morning of every treatment day of the adriamycin/cytoxan cycles; they will receive acupuncture for every third Taxol treatment, beginning with the first treatment. They will receive a total of 8 acupuncture sessions: 4 with the adriamycin/cytoxan cycles and 4 with the Taxol cycles. Both groups will fill out MDASI on day 3 (+/- 1 days) of each Adriamycin/Cytoxan cycle; they will also fill out the MDASI on day 3 (+/- 1 days) of every third Taxol treatment for a total of 8 MDASI forms.
- Chemotherapy 3 No Acupuncture (No Intervention): Chemotherapy 3: In the adjuvant setting- This group will receive Taxotere (75mg/m2) and Cytoxan (600 mg/m2) on day 1 every 3 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Cytoxan for a total of 4 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 4 MDASI forms.
- Chemotherapy 4 No Acupuncture (No Intervention): Chemotherapy 4: In the neoadjuvant setting- This group will receive Taxotere (75 mg/m2), Carboplatin (AUC 6), Perjeta (840 mg loading fixed dose, followed by 420 mg maintenance fixed dose) day 1 every 3 weeks for 6 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Carboplatin/Perjeta treatment for a total of 6 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 6 MDASI forms.

INTERVENTIONS:
Device: Acupuncture
  Arms: Chemotherapy 1 Acupuncture; Chemotherapy 2 Acupuncture; Chemotherapy 3 Acupuncture; Chemotherapy 4 Acupuncture

SUMMARY:
The goal of this study is to determine if acupuncture improves multiple symptoms associated with chemotherapy on the MD Anderson Symptom Inventory (MDASI): nausea, vomiting, fatigue, anxiety, anorexia, pain, disturbed sleep, shortness of breath, dry mouth, depression, and peripheral neuropathy (see statistical section). The investigators hypothesis is that acupuncture will result in lower MDASI scores over the course of chemotherapy for the acupuncture group vs. control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking/reading/writing
* Breast cancer stages I through III
* Any performance status suitable for chemotherapy as determined by the physician
* Primary or secondary chemotherapy, but enrolling patients prior to a chemotherapy regimen regardless of previous radiation therapy exposure and/or previous mastectomy.
* Scheduled to receive either of the following two regimens:
* Adriamycin (60 mg/m2), Cytoxan (600 mg/m2), Taxol (175 mg/m2)
* Adriamycin (60 mg/m2), Cytoxan (600 mg/m2), Taxol (80 g/m2)
* Taxotere (75mg/m2), Cytoxan (600 mg/m2)
* Taxotere (75 mg/m2), Carboplatin (AUC 6), Perjeta (840 mg loading fixed dose, followed by 420 mg maintenance fixed dose)

Exclusion Criteria:

* History of narcolepsy
* Sleep apnea requiring continuous positive airway pressure (CPAP)
* Other acupuncture treatment within one month of enrollment
* Acupuncture treatment for chemotherapy in the past
* Current participation in any other research studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Bell, MD, Principal Investigator — OhioHealth
Locations (1):
- Columbus Oncology and Hematology Associates, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy 1 Acupuncture; Chemotherapy 1 No Acupuncture: Chemotherapy 1: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) concurrently on day 1 every 2 weeks for 4 cycles followed by Taxol (175mg/m2) on day 1 every 2 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every treatment for a total of 8 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 8 MDASI forms.
  Acupuncture
  No Acupuncture- Standard of Care
- Chemotherapy 2 Acupuncture; Chemotherapy 2 No Acupuncture: Chemotherapy 2: This group will receive Adriamycin (60mg/m2) and Cytoxan (600mg/m2) on day 1 every 2 weeks for 4 cycles followed by Taxol (80mg/m2) on day 1 weekly for 12 cycles. Patients who randomize to the experimental ("acupuncture") group will undergo acupuncture the morning of every treatment day of the adriamycin/cytoxan cycles; they will receive acupuncture for every third Taxol treatment, beginning with the first treatment. They will receive a total of 8 acupuncture sessions: 4 with the adriamycin/cytoxan cycles and 4 with the Taxol cycles. Both groups will fill out MDASI on day 3 (+/- 1 days) of each Adriamycin/Cytoxan cycle; they will also fill out the MDASI on day 3 (+/- 1 days) of every third Taxol treatment for a total of 8 MDASI forms.
  Acupuncture
  No Acupuncture- Standard of Care
- Chemotherapy 3 Acupuncture; Chemotherapy 3 No Acupuncture: Chemotherapy 3: In the adjuvant setting- This group will receive Taxotere (75mg/m2) and Cytoxan (600 mg/m2) on day 1 every 3 weeks for 4 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Cytoxan for a total of 4 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 4 MDASI forms.
  Acupuncture
  No Acupuncture- Standard of Care
- Chemotherapy 4 Acupuncture; Chemotherapy 4 No Acupuncture: Chemotherapy 4: In the neoadjuvant setting- This group will receive Taxotere (75 mg/m2), Carboplatin (AUC 6), Perjeta (840 mg loading fixed dose, followed by 420 mg maintenance fixed dose) day 1 every 3 weeks for 6 cycles. Patients on this regimen who randomize to the experimental ("acupuncture") group will undergo acupuncture on the morning of every Taxotere/Carboplatin/Perjeta treatment for a total of 6 acupuncture sessions. Both groups will complete a MDASI on day 3 (+/- 1 days) of each cycle of chemotherapy for a total of 6 MDASI forms.
  Acupuncture
  No Acupuncture- Standard of Care
Period: Overall Study
Arm/Group | Chemotherapy 1 Acupuncture | Chemotherapy 2 Acupuncture | Chemotherapy 3 Acupuncture | Chemotherapy 4 Acupuncture | Chemotherapy 1 No Acupuncture | Chemotherapy 2 No Acupuncture | Chemotherapy 3 No Acupuncture | Chemotherapy 4 No Acupuncture
Started | 3 | 3 | 0 | 0 | 2 | 2 | 0 | 0
Completed | 3 | 3 | 0 | 0 | 2 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy 1 Acupuncture | Chemotherapy 2 Acupuncture | Chemotherapy 3 Acupuncture | Chemotherapy 4 Acupuncture | Chemotherapy 1 No Acupuncture | Chemotherapy 2 No Acupuncture | Chemotherapy 3 No Acupuncture | Chemotherapy 4 No Acupuncture | Total
Number analyzed (Participants) | 3 | 3 | 0 | 0 | 2 | 2 | 0 | 0 | 10
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  |  | 0 | 0 |  |  | 0
  Between 18 and 65 years | 1 | 3 |  |  | 2 | 2 |  |  | 8
  >=65 years | 2 | 0 |  |  | 0 | 0 |  |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (15.7) | 43.2 (12.0) |  |  | 45.0 (14.9) | 49.0 (18.1) |  |  | 50.1 (13.5)
Gender [Number; unit: participants]
  Female | 3 | 3 |  |  | 2 | 2 |  |  | 10
  Male | 0 | 0 |  |  | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 |  |  | 2 | 2 |  |  | 10

OUTCOME MEASURES:

1. Primary Outcome: MDASI Score of Chemotherapy-associated Symptoms With Acupuncture Treatment
Description: The investigators will first plot M.D. Anderson Symptom Inventory Core Items (MDASI) scores over time for the acupuncture and control groups to visually inspect for differences between the two groups. The investigators will further evaluate the difference in MDASI scores for the two groups using linear mixed models that account for multiple measurements within a single patient. A mixed model is preferable to a repeated measures ANOVA in this case, as it allows for missing time points within a single subject without eliminating that subject from the analysis.
  Additionally, the investigators are able to specify how our time points are correlated within patients rather than assuming equal correlation across time points. The MDASI is comprised of 13 separate items that are not summative; therefore, the significance level for all statistical tests will be set at 0.003 (0.05/13) to account for multiple comparisons.
Time Frame: 15 months
Population: Per IRB guidelines, we were not permitted to analyze the 10 patients enrolled since we did not meet completed enrollment numbers.
Arm/Group | Acupuncture | Standard of Care- No Acupuncture
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy 1 Acupuncture | Chemotherapy 1 No Acupuncture | Chemotherapy 2 Acupuncture | Chemotherapy 2 No Acupuncture | Chemotherapy 3 Acupuncture | Chemotherapy 3 No Acupuncture | Chemotherapy 4 Acupuncture | Chemotherapy 4 No Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/2 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/3 | 0/2 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No